CLINICAL TRIAL: NCT02562950
Title: A Phase I, Open Interaction Study Between Oral Doses of GLPG1837 and Single Doses of Midazolam in Healthy Male Subjects
Brief Title: A Phase I, Open Interaction Study Between GLPG1837 and Midazolam in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1837-CL-102; 2015-002517-29 (EudraCT Number)
Record Dates: First submitted 2015-09-23; First posted 2015-09-29 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1837; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam and 500 mg GLPG1837 (Experimental): Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions (Days 1 and 12) and multiple oral doses of GLPG1837 (250 mg b.i.d daily for 10 days) from Days 2 to 11.
  Interventions: Drug: GLPG1837 500 mg; Drug: Midazolam
- Midazolam and 1000 mg GLPG1837 (Experimental): Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions (Days 1 and 12) and multiple oral doses of GLPG1837 (500 mg b.i.d daily for 11 days) from Days 2 to 12.
  Interventions: Drug: Midazolam; Drug: GLPG1837 1000 mg

INTERVENTIONS:
Drug: GLPG1837 500 mg — Each subject will receive multiple oral daily doses of GLPG1837 (250 mg b.i.d. for 11 days) from Days 2 to 12.
  Arms: Midazolam and 500 mg GLPG1837
Drug: Midazolam — Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions (Days 1 and 12).
Drug: GLPG1837 1000 mg — Each subject will receive multiple oral doses of GLPG1837 (500 mg b.i.d. for 11 days) from Days 2 to 12.
  Arms: Midazolam and 1000 mg GLPG1837

SUMMARY:
This will be a drug-drug interaction study to evaluate the effect of multiple oral doses of GLPG1837 on the single dose pharmacokinetic profile of midazolam administered in fed healthy male subjects. Each subject will receive a single oral dose of midazolam (2 mg) on 2 occasions: on Day 1, before dosing with GLPG1837 and on Day 12 co-administered with GLPG1837, after multiple oral doses of GLPG1837 (daily for 10 days, from Day 2 until Day 11).

Also, the safety and tolerability of multiple oral doses of GLPG1837 co-administered with midazolam in healthy male subjects will be evaluated.

A first dose group of 12 subjects will receive a total daily dose of 500 mg (250 mg b.i.d.) GLPG1837 and a second dose group of 12 subjects will receive a total daily dose of 1000 mg (500 mg b.i.d.) GLPG1837.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The maximum observed concentration (Cmax) of (1'-OH) Midazolam in plasma before and after multiple oral doses of GLPG1837 | Between Day 1 (predose) and Day 13 (24h post last dose on Day 12)
  To characterize the maximum observed concentration (Cmax) of (1'-OH) Midazolam in plasma over time before and after multiple doses of GLPG1837 in healthy male subjects
The time of occurrence of Cmax (tmax) of (1'-OH) Midazolam in plasma before and after multiple oral doses of GLPG1837 | Between Day 1 (predose) and Day 13 (24h post last dose on Day 12)
  To characterize the time of occurrence of Cmax (tmax) of (1'-OH) Midazolam in plasma before and after multiple doses of GLPG1837 in healthy male subjects
The area under the plasma concentration versus time curve (AUC) of (1'-OH) Midazolam before and after multiple oral doses of GLPG1837 | Between Day 1 (predose) and Day 13 (24h post last dose on Day 12)
  To characterize the area under the plasma concentration versus time curve (AUC) of (1'-OH) Midazolam before and after multiple doses of GLPG1837 in healthy male subjects
The apparent terminal half-life (t1/2) of (1'-OH) Midazolam in plasma before and after multiple oral doses of GLPG1837 | Between Day 1 (predose) and Day 13 (24h post last dose on Day 12)
  To characterize the apparent terminal half-life (t1/2) of (1'-OH) Midazolam in plasma before and after multiple doses of GLPG1837 in healthy male subjects

SECONDARY OUTCOMES:
The maximum observed concentration (Cmax) of GLPG1837 (metabolite) in plasma after multiple oral doses of GLPG1837 (and co-administration of Midazolam on Day 12) | Between Day 5 (predose) and Day 14 (48h after the last dose on Day 12)
  To characterize the maximum observed concentration (Cmax) of GLPG1837 (metabolite) in plasma after multiple doses of GLPG1837 (and co-administration of Midazolam on Day 12) in healthy male subjects
Number of adverse events | Between Screening and 7-10 days after the last dose of GLPG1837 on Day 12
  To evaluate the safety and tolerability of GLPG1837 after multiple oral doses in healthy male subjects with or without coadministration of Midazolam in terms of the number of adverse events reported
Changes in vital signs as measured by heart rate, blood pressure, respiratory rate and oral body temperature | Between Screening and 7-10 days after the last dose of GLPG1837 on Day 12
  To evaluate the safety and tolerability of GLPG1837 after multiple oral doses in healthy male subjects with or without coadministration of Midazolam in terms of changes in vital signs as measured by heart rate, blood pressure, respiratory rate and oral body temperature reported
Changes in 12-lead ECG measures | Between Screening and 7-10 days after the last dose of GLPG1837 on Day 12
  To evaluate the safety and tolerability of GLPG1837 after multiple oral doses in healthy male subjects with or without coadministration of Midazolam in terms of changes in 12-ECG measures reported
Changes in physical exam measures | Between Screening and 7-10 days after the last dose of GLPG1837 on Day 12
  To evaluate the safety and tolerability of GLPG1837 after multiple oral doses in healthy male subjects with or without coadministration of Midazolam in terms of changes in physical examination reported
Changes in blood safety lab parameters | Between Screening and 7-10 days after the last dose of GLPG1837 on Day 12
  To evaluate the safety and tolerability of GLPG1837 after multiple oral doses in healthy male subjects with or without coadministration of Midazolam in terms of changes in blood safety lab parameters reported
Changes in urine safety lab parameters | Between Screening and 7-10 days after the last dose of GLPG1837 on Day 12
  To evaluate the safety and tolerability of GLPG1837 after multiple oral doses in healthy male subjects with or without coadministration of Midazolam in terms of changes in urine safety lab parameters reported
The time of occurrence of Cmax (tmax) of GLPG1837 (metabolite) in plasma after multiple oral doses of GLPG1837 (and co-administration of Midazolam on Day 12) | Between Day 5 (predose) and Day 14 (48h after the last dose on Day 12)
  To characterize the time of occurrence of Cmax (tmax) of GLPG1837 (metabolite) in plasma after multiple doses of GLPG1837 (and co-administration of Midazolam on Day 12) in healthy male subjects
The area under the plasma concentration versus time curve (AUC) of GLPG1837 (metabolite) in plasma after multiple oral doses of GLPG1837 (and co-administration of Midazolam on Day 12) | Between Day 5 (predose) and Day 14 (48h after the last dose on Day 12)
  To characterize the area under the plasma concentration versus time curve (AUC) of GLPG1837 (metabolite) in plasma after multiple doses of GLPG1837 (and co-administration of Midazolam on Day 12) in healthy male subjects
The apparent terminal half-life (t1/2) of GLPG1837 (metabolite) in plasma after multiple oral doses of GLPG1837 (and co-administration of Midazolam on Day 12) | Between Day 5 (predose) and Day 14 (48h after the last dose on Day 12)
  To characterize the apparent terminal half-life (t1/2) of GLPG1837 (metabolite) in plasma after multiple doses of GLPG1837 (and co-administration of Midazolam on Day 12) in healthy male subjects
The metabolite to GLPG1837 ratios in plasma after multiple oral doses of GLPG1837 (and co-administration of Midazolam on Day 12) | Between Day 5 (predose) and Day 14 (48h after the last dose on Day 12)
  To characterize the metabolite to GLPG1837 ratios in plasma after multiple doses of GLPG1837 (and co-administration of Midazolam on Day 12) in healthy male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium